CLINICAL TRIAL: NCT01844271
Title: Low Level Laser Therapy in Muscle Fatigue and Muscle Recovery After Exercise: What is the Ideal Dose?
Brief Title: Low Level Laser Therapy in Muscle Fatigue and Muscle Recovery
Acronym: LLLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Adriane Aver Vanin, Low level laser therapy in muscle fatigue and muscle recovery after exercise: what is the ideal dose?, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Uninove
Record Dates: First submitted 2013-04-24; First posted 2013-05-01 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Muscle; Fatigue, Heart; Skeletal Muscle Recovery
Keywords: LLLT; muscle fatigue and recovery; phototherapy parameter
MeSH Terms: conditions — Fatigue | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo Low Level Laser (Placebo Comparator): Application of low level laser without any dose (0 Joule) before strenuous exercise. A laser device with a cluster of 5 diodes (810 nm, 200 mW) each diode was used for this study.
  Interventions: Device: Low Level Laser (LLL)
- 2 Joules Low Level Laser (Experimental): Application of 2 Joules of Low Level Laser Therapy before strenuous exercise with a cluster of 5 diode (810 nm, 200 mW each diode).
  Interventions: Device: Low Level Laser (LLL)
- 6 Joules Low Level Laser Therapy (Experimental): Application of 6 Joules of Low Level Laser Therapy before strenuous exercise with a cluster of 5 diode (810 nm, 200 mW each diode).
  Interventions: Device: Low Level Laser (LLL)
- 10 Joules Low Level Therapy (Experimental): Application of 10 Joules of Low Level Laser Therapy before strenuous exercise with a cluster of 5 diode (810 nm, 200 mW each diode).
  Interventions: Device: Low Level Laser (LLL)
- Power of 100mW (Experimental): After assigning ideal dose of application it was delimited two experimental groups which was irradiated with the dose established by the first part of the study and power of 100mW.
  Interventions: Device: Low Level Laser (LLL)
- Power of 400mW (Experimental): After assigning ideal dose of application it was delimited two experimental groups which were irradiated with the dose established by the first part of the study and power of 400mW.
  Interventions: Device: Low Level Laser (LLL)

INTERVENTIONS:
Device: Low Level Laser (LLL) — Comparison of different dosages of a Low Level Laser applied in six different locations of the knee extensor muscles of the lower limb non-dominant before a strenuous exercise.
  We performed stretching and warming up of the muscles involved, assessment of muscle pain, withdrawal of blood sample, test muscle function (MVC), application of dose of low level laser designated for each volunteer (0, 2, 6 or 10), performing eccentric contractions protocol in isokinetic dynamometer . After the protocol we evaluated muscle function, the DOMS, and blood analyzes in 1 minute, 1 hour, 24 hours, 48 hours 72 hours and 96 hours.
  In a second stage, the optimal dose defined by the first part of the study will be tested in two different powers, 100 and 400mW. The study was repeated in two experimental groups using the optimal dose established and the powers of 100 and 400mW that was randomly distributed in groups.

SUMMARY:
Muscle fatigue and muscle recovery after exercise are recent areas of research involving Low Level Laser Therapy (LLLT) and many factors remain unknown, such as optimal doses, power and application parameters, mechanisms of action, effects on long-term exercise and the long-term effects on skeletal muscle recovery.

The present research project aims to assess the effects of long-term recovery of LLLT in skeletal muscle after exercise and identify the optimal dose application of LLLT.

After defining the best dose of application, we recruited two groups which will be irradiated with different power, 100mW and 400mW in order to seek the optimal parameter of low level laser therapy in performance.

The investigators believed that the Low Level Laser Therapy can delay the physiological process of muscle fatigue, reduce injury or skeletal muscle microdamage arising from physical effort and accelerate muscle recovery after exercise.

DETAILED DESCRIPTION:
To achieve the proposed objectives it was performed a randomized, double-blinded, placebo-controlled trial, with voluntary participation of high-level soccer athletes.

Participants received an application of low level laser prior to execution of a strenuous exercise. It was used a laser with a cluster of 5 diodes (810 nm, 200 mW each diode) with different doses (placebo, 2J, 6J, 10J) and power of 200mW.

In a second step, with the optimal dose already defined, this was used to be applied with different powers in two experimental groups, 100mW and 400mW.

The investigators analysed parameters related to volunteers exercise performance (torque peak / maximum voluntary contraction), delayed onset muscle soreness, and biochemical markers of muscle damage (CK and LDH), inflammation (interleukin 1 and 6, alpha tumoral necrosis factor) and oxidative stress (TBARS, CAT, SOD and carbonylated proteins). The analysis was performed before exercise protocols, after 1 minute, and 1, 24, 48, 72 and 96 hours after the end of exercise protocol in both parts of the study.

ELIGIBILITY:
Inclusion Criteria:

* professional soccer players aged between 18 and 35 years old;
* not presenting historical musculoskeletal injury in regions of the hip and knee in the 2 months preceding the study;
* not making use of pharmacological agents and/or nutritional supplements;
* participating with minimum frequency of 80% of the training team

Exclusion Criteria:

* athletes who experience musculoskeletal injury during the study;
* athletes who for whatever reason have their training routine changed with respect to the rest of the team during the course of study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-05; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Exercise performance (MVC and peak torque) | Maximum voluntary contraction (MVC) was performed before the exercise protocol and repeted 1 minute, 1 hour, 24, 48, 72 and 96 hours after the eccentric contraction protocol. The peak torque was performed after 3 minutes of LLLT application.
  The investigators used an isokinetic dynamometer to assess muscle function and the execution of the exercise protocol, because this tool is currently recognized as the most reliable, reliability and reproducibility for measuring the performance musculoskeletal.
  The maximum voluntary contraction (MVC) was performed before the exercise protocol and repeated 1 minute, 1 hour, 24, 48, 72 and 96 hours after the eccentric contraction protocol.
  The peak torque was measured after evaluation of muscular pain, blood tests, stretching and warming, MVC and application of a predetermined dose of low level therapy (LLLT). It was done after 3 minutes of LLLT application through execution of a eccentric contraction of 5 series of 15 repetitions.
  After the execution of the exercise protocol it was repeated the collection of blood samples, measuring DOMS and muscle function test (MVC) in 1 minute, 1 hour, 24 hours, 48 hours, 72 hours and 96 hours from the protocol.

SECONDARY OUTCOMES:
Blood tests (composite measures) | Analysis of biochemical markers of muscle damage, inflammation and oxidative stress before exercise protocols, after 1 minute, and 1, 24, 48, 72 and 96 hours after the end of exercise protocol.
  Biochemical markers of muscle damage (CK and LDH), inflammation (IL-1, IL-6 and tumor necrosis factor(TNF)-alpha) and oxidative stress (TBARS, CAT, SOD and carbonylated proteins). The analysis were performed before exercise protocols, after 1 minute, and 1, 24, 48, 72 and 96 hours after the end of exercise protocol.

OTHER OUTCOMES:
Delayed onset muscle soreness (DOMS) | The analysis were performed before exercise protocols, after 1 minute, and 1, 24, 48, 72 and 96 hours after the end of exercise protocol.
  Assessed through an analog algometer always by the same investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Adriane A Vanin, PT, Study Chair — Nove de Julho University
Locations (1):
- Nove de Julho University, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Baroni BM, Leal Junior EC, De Marchi T, Lopes AL, Salvador M, Vaz MA. Low level laser therapy before eccentric exercise reduces muscle damage markers in humans. Eur J Appl Physiol. 2010 Nov;110(4):789-96. doi: 10.1007/s00421-010-1562-z. Epub 2010 Jul 3. PMID 20602109
- [Derived] de Oliveira AR, Vanin AA, De Marchi T, Antonialli FC, Grandinetti Vdos S, de Paiva PR, Albuquerque Pontes GM, Santos LA, Aleixo Junior Ide O, de Carvalho Pde T, Bjordal JM, Leal-Junior EC. What is the ideal dose and power output of low-level laser therapy (810 nm) on muscle performance and post-exercise recovery? Study protocol for a double-blind, randomized, placebo-controlled trial. Trials. 2014 Feb 27;15:69. doi: 10.1186/1745-6215-15-69. PMID 24576321